CLINICAL TRIAL: NCT05887648
Title: Effect of Singapore-contextualized Dance-based Exergame (SinDance) in Promoting Physical Function and Reducing Depressive Symptoms and Falls Among Community-dwelling Older Adults: A Randomised Controlled Trial
Brief Title: Effect of Singapore-contextualized Dance-based Exergame Among Community-dwelling Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Collaborators: National University Hospital, Singapore (Other); Lions Befrienders Service Association (Singapore) (Unknown)
Responsible Party: Principal Investigator, Jiang Ying, Assistant Professor, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NUHS Seed Grant Call Sep 2021
Record Dates: First submitted 2023-05-09; First posted 2023-06-05 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Community-dwelling Older Adults
Keywords: falls; activities of daily living; exercise; dance; exergame
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants are randomised into 2 groups - SinDance (interventional group) or control group. A computerised randomisation programme will generate the randomization list and a person independent from the study will prepare the sealed envelopes according to the generated randomisation list. After a participant is registered, a unique participant enrolment ID will be assigned to the participant. The envelope according to the enrolment ID will be opened on site and the participant will be allocated into either one of the two groups based on the randomisation list the group indicated.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SinDance (Experimental): Participants in the SinDance group will attend an educational briefing session on the importance of exercising, and participate in a 6-week SinDance exergame intervention
  Interventions: Behavioral: SinDance
- Control (No Intervention): Participants in the control group will attend usual activities offered by the senior activity centres. The control group will be offered an opportunity to play the SinDance exergame after completing the last data collection (i.e. 3-months from baseline).

INTERVENTIONS:
Behavioral: SinDance — One face-to-face briefing session (20 min) will be offered to participants in the SinDance group as part of promoting physical activity and safe exercise for older adults.
  Participants will be asked to engage in SinDance 3 times a week for 6 weeks. Each session will last for about 30-40 mins, including 5 mins warm up exercise before the game and 5 mins cool down exercise afterwards.
  All the game play sessions will be conducted in LB centres. Each participant will play the game individually.
  To play the game, participants will dance to the dance moves shown on the screen (on the external monitor or the projected screen) and as they get each move right, they will be awarded points. The more accurate their moves are, the more points they get in the game.
  During the gameplay, the participants will be instructed to stop and rest if they are tired. A RN/RA will be on site to observe the safety of exergaming and to help resolve technical issues as they arise.
  Arms: SinDance

SUMMARY:
The aims of the research are to develop an age-appropriate and culturally sensitive older person-centered, Singapore-contextualized Dance-based Exergame (SinDance), and to pilot test its effectiveness in improving physical function and activity daily living (ADL) and reducing depressive symptoms and falls among community-dwelling older people. It is hypothesized that participants in the SinDance will have: (1) improved postural balance, muscle strength, and ADL; and (2) reduced depressive symptoms, fear of falling, and number of falls, compared to those in the control group.

The research will be structured as a two-phase study.

1. In Phase one, development of the SinDance system will be undertaken.
2. In Phase two, a pilot randomized control trial will be conducted to evaluate the feasibility and potential effectiveness of the newly developed SinDance exergame on the proposed outcomes.

   * Eligible participants will be recruited from Lions Befrienders (LB) senior activity centre and randomly assigned to the SinDance group or the control group.
   * Participants in the intervention group will receive one face-to-face briefing session and will be required to participate in the newly developed SinDance exergame 3 times a week for 6 weeks, while those in the control group will attend usual activities provided by the centers.
   * Outcomes will be measured at baseline, immediate after intervention, and 3 months from baseline.

DETAILED DESCRIPTION:
SinDance will be structured as a two-phase study involving a multi-disciplinary team of software engineers, occupational therapist (OT), and research nurse (RN).

Phase 1: Development of the SinDance system will be undertaken by software engineers in collaboration with an OT and RN.

* The SinDance intervention is a 6-week program consisting of one face-to-face briefing session provided by the Research Nurse (RN)/Research Assistant (RA) and SinDance exergaming. The dance movements will be choreographed for older adults based on local context and culture. The game design of SinDance will be developed on cross-platform game engine called Unity. Body movements will be captured via an external RGB camera. Using an open pose algorithm, the system will be able to track correct body movements based on image processing and body posture recognition, as well as provide active feedback on performance. This allows for real-time movement adjustments by the user to achieve higher compliance rating. Points will be awarded for each correct movement accomplished.
* The SinDance intervention is designed as a leisure game to supplement the daily physical activities of older adults. There will NOT be strenuous or intense physical activities or any vigorous high-velocity movements in this intervention.

Considering that SinDance is a self-regulated exercise, to ensure safety during self-regulated exercise, dance choreography will be designed with varying levels of movement difficulty, speed and rhythm tempo to cater to the different needs of individual participants. The SinDance game interface will be designed with minimal action buttons to enhance usability and user- experience for older people to operate.

Phase 2: Pilot test to assess the effectiveness of SinDance exergame Study Design - A pilot two-arm randomized control trial with repeated measures will be conducted in Phase 2. Eligible participants will be recruited from Lions Befrienders (LB) senior activity centre. They will be randomly allocated to either intervention group or control group using block randomisation technique. The data will be collected at baseline, immediately after the intervention (i.e., 6 weeks from baseline) and 3 months from baseline.

Study Intervention

* The exergame will run on a laptop, the display of game will be either on an external monitor or project to screen via a projector. To play the game, participants will dance to the dance moves shown on the screen and as they get each move right, they will be awarded points (please see attached picture for the proposed interface design and system setup). The RGB webcams will be used to capture body movements and provide immediate/spontaneous feedback on the correctness of the movements. It will be affixed to the laptop. The participants' faces will not be captured.
* There will be no device for the participants to take home. The participants will only play the game in LB SACs (not in their homes).
* For this study, the participant will play the game individually, and under the observation of a RA/RN to ensure safety. No group play will be conducted in the pilot study. Before playing, they will be briefed on how to play in a language they understand.

SinDance Group.

* One face-to-face briefing session will be offered to participants in the SinDance group. The session will be conducted by the RN/RA. As part of promoting physical activity and safe exercise for older adults, the RN/RA will provide general guidance to older people on the benefits of physical activity (e.g.the recommended duration for physical activity, which will yield health benefits, and therefore, participants will play the exergame for 3 times a week and each session about 30 mins) and how to exercise safely (e.g. don't exercise if you feel unwell or very tired, wear appropriate footwear, warm up before exercise and cool down and stretch after exercise, etc.). This education will be provided to intervention group only. He/She will also teach the participants on how to navigate the SinDance exergame system, and how to choose between different levels of dance and play modes. It is estimated that the session will last for 20 minutes.
* To achieve adequate exercise volume, participants will be asked to engage in the newly developed SinDance 3 times a week for 6 weeks. Each session will last for about 30-40 mins, including 5 mins warm up exercise before the game and 5 mins cool down exercise afterwards. Therefore, if the participant does not stop halfway through or end the game early, the actual playing time for each participant will be about 20-30 minutes.
* To play the game, participants will dance to the dance moves shown on the screen (on the external monitor or the projected screen) and as they get each move right, they will be awarded points. The more accurate their moves are, the more points they get in the game.
* During the gameplay, the participants will be instructed to stop and rest if they are tired, and to dance on their own without the physical assistance from others during their play. A RN/RA will be on site to observe the safety of exergaming and to help resolve technical issues as they arise.

Control Group.

- Participants in the control group will attend usual activities offered by the senior activity centres. The control group will be offered an opportunity to play the SinDance exergame after completing the last data collection (i.e. 3-months from baseline).

ELIGIBILITY:
Inclusion Criteria:

1. Age 60 and above
2. Living in the community
3. Independent without use of walking aids
4. able to read and understand English or Chinese
5. TUG < 30s
6. Mini-Cog test score of 3 and above

Exclusion Criteria:

1. Are suffering from mental disorders or cognitive impairment that will prevent individuals from understanding the study and performing the exergame correctly and safely (e.g. Alzheimer's disease)

   - Mini-Cog less than 3
2. have a pre-existing medical condition that prohibits exercise, or prevents the individual from performing the exergame correctly and safely, including but not limited to:

   * chest pain or chest tightness during physical activities (e.g. walking, climbing stairs, doing household chores or similar activities
   * heart failure
   * currently experience dizziness or light-headedness, uncontrolled/unstable high blood pressure
3. have physical limitations, for examples:

   * wheelchair bound
   * pain, stiffness or swelling that will prevent the individual from doing what he/she wants or need to do
   * feel unsteady, use an assistive device while standing or walking
   * TUG equal or more than 30 seconds
4. have visual or hearing impairments.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-04-05 (Actual); Primary Completion 2024-01-24 (Actual); Study Completion 2024-01-24 (Actual)

PRIMARY OUTCOMES:
Short Fall Efficacy Scale International (short FES-I) | Baseline
  Scores range from 7 to 28 and lower scores indicate a better outcome (lower fear of falling).
Short Fall Efficacy Scale International (short FES-I) | 6 weeks from baseline
  Scores range from 7 to 28 and lower scores indicate a better outcome (lower fear of falling).
Short Fall Efficacy Scale International (short FES-I) | 3 months from baseline
  Scores range from 7 to 28 and lower scores indicate a better outcome (lower fear of falling).
15-item Geriatric Depression Scale (GDS-15) | Baseline
  Scores range from 0-15, and higher scores indicate a worse outcome (depression).
15-item Geriatric Depression Scale (GDS-15) | 6 weeks from baseline
  Scores range from 0-15, and higher scores indicate a worse outcome (depression).
15-item Geriatric Depression Scale (GDS-15) | 3 months from baseline
  Scores range from 0-15, and higher scores indicate a worse outcome (depression).
Frenchay Activities Index (FAI) | Baseline
  Scores range from 15-60 and higher scores indicate better outcome (better ability to engage in activities of daily living)
Frenchay Activities Index (FAI) | 6 weeks from baseline
  Scores range from 15-60 and higher scores indicate better outcome (better ability to engage in activities of daily living)
Frenchay Activities Index (FAI) | 3 months from baseline
  Scores range from 15-60 and higher scores indicate better outcome (better ability to engage in activities of daily living)
Five times sit-to-stand test (FTSTS) | Baseline
  A longer time taken to complete the test indicates a worse outcome (weaker functional lower limb muscle strength)
Five times sit-to-stand test (FTSTS) | 6 weeks from baseline
  A longer time taken to complete the test indicates a worse outcome (weaker functional lower limb muscle strength)
Five times sit-to-stand test (FTSTS) | 3 months from baseline
  A longer time taken to complete the test indicates a worse outcome (weaker functional lower limb muscle strength)
Time Up & Go Test (TUG) | Baseline
  A longer time to complete the test indicates a worse outcome (poorer mobility)
Time Up & Go Test (TUG) | 6 weeks from baseline
  A longer time to complete the test indicates a worse outcome (poorer mobility)
Time Up & Go Test (TUG) | 3 months from baseline
  A longer time to complete the test indicates a worse outcome (poorer mobility)
Functional Reach Test | Baseline
  A longer reach distance indicates a better outcome (better balance)
Functional Reach Test | 6 weeks from baseline
  A longer reach distance indicates a better outcome (better balance)
Functional Reach Test | 3 months from baseline
  A longer reach distance indicates a better outcome (better balance)
Modified Barthel ADL Index | Baseline
  Scores range from 0-20, and higher scores indicate a better outcome (functional independence in the domains of personal care and mobility)
Modified Barthel ADL Index | 6 weeks from baseline
  Scores range from 0-20, and higher scores indicate a better outcome (functional independence in the domains of personal care and mobility)
Modified Barthel ADL Index | 3 months from baseline
  Scores range from 0-20, and higher scores indicate a better outcome (functional independence in the domains of personal care and mobility)

SECONDARY OUTCOMES:
Attendance (for SinDance group only) | Each session during the 6-week intervention (total of 18 sessions)
  Their attendance for each exergame session will be recorded
Level of motivation (for SinDance group only) | Each session during the 6-week intervention (total of 18 sessions)
  Participants will be asked to rate their level of motivation to play the exergame after each exergame session on a five-point Likert scale ranging from '1 = very low' to '5 = very high'.
Level of enjoyment (for SinDance group only) | Each session during the 6-week intervention (total of 18 sessions)
  Participants will be asked to rate their level of enjoyment during the exergame after each exergame session on a five-point Likert scale ranging from '1 = very low' to '5 = very high'.
Duration of play (for SinDance group only) | Each session during the 6 week intervention (total of 18 sessions)
  Their duration of play for each exergame session will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Ying Jiang, PhD, Principal Investigator — Alice Lee Centre for Nursing Studies, National University of Singapore
Locations (5):
- Singapore (5):
  - Lions Befrienders Active Ageing Centre @ CLEMENTI 344, Singapore
  - Lions Befrienders Active Ageing Centre @ CLEMENTI 366/367, Singapore
  - Lions Befrienders Active Ageing Centre @ CLEMENTI 420A, Singapore
  - Lions Befrienders Active Ageing Centre @ Bendemeer 32, Singapore
  - Lions Befrienders Active Ageing Centre @ Tampines 499C, Singapore

IPD SHARING:
Plan to Share IPD: Yes
Anonymised study results and data will be available to researchers who request it as part of an IPD study or meta-analysis that has been prospectively registered and a protocol by a representative researcher is provided to verify the legitimacy of the request.
Supporting Information: ICF
Time Frame: Data will be available following publication of the study's results in a peer-reviewed journal
Access Criteria: Anonymised study results and data will be available to researchers who request it as part of an IPD study or meta-analysis that has been prospectively registered and a protocol by a representative researcher is provided to verify the legitimacy of the request.